CLINICAL TRIAL: NCT02723396
Title: Sleep & Move. Systematic Characterisation of Sleep Benefit in Parkinson's Disease. An Observational, Prospective Study
Brief Title: Sleep, Awake & Move - Part I
Acronym: SA&M-I
Status: Completed | Type: Observational
Sponsor: Neurocenter of Southern Switzerland (Other)
Collaborators: Parkinson Schweiz (Other); Ente Ospedaliero Cantonale, Bellinzona (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Pietro Luca Ratti, MD, PhD, Neurocenter of Southern Switzerland
Other Study IDs: EOC.NSI.LS.15.3.I
Record Dates: First submitted 2016-03-12; First posted 2016-03-30 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Parkinson Disease
Keywords: Parkinson's disease; Sleep Benefit
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson: Prospective observation of a cohort of consecutive patients with idiopathic PD in an ecological setting.
- Healthy: The same assessments will be performed in a subgroup of age- and sex-matched healthy volunteers.

SUMMARY:
Sleep benefit (SB) is a prominent spontaneous, apparently unpredictable, transitory improvement in motor function reported by around 50% of patients affected by Parkinson's Disease (PD) after sleep and before taking their first dose of dopaminergic medications. This study aims at systematically characterizing SB in PD patients in an ecological setting and to explore the relationships between nocturnal and diurnal sleep and subjective and objective measures of motor function. A better understanding of this phenomenon is mandatory for future research on this topic.

DETAILED DESCRIPTION:
The "Sleep & Move" study is the first part of the Sleep, Awake & Move project. In this observational study we plan to systematically investigate SB and the day-to-day variation in this phenomenon in PD patients by a prospective, repeated assessment for 14 days of both subjective and objective measures of motor function and sleep at patients' home, by an Android app developed ad hoc by our group and named "SleepFit".

Since is still unknown if a spontaneous, subclinical improvement in motor performance might also occur in healthy subjects or if the SB is a phenomenon only involving subjects with PD, we had the idea to test this hypothesis comparing a subgroup of PD patients with age- and sex-matched healthy volunteers, employing the same assessments as in the Sleep & Move study.

ELIGIBILITY:
PARKINSON'S DISEASE GROUP:

Inclusion Criteria:

* Diagnostic criteria of idiopathic Parkinson's disease (UKPDBB)
* Mild to moderate disease (Hoehn & Yahr score ≥ 1 and <= 3)
* Mentally and physically capable to give informed consent
* Stable antiparkinsonian and psychotropic therapy for the last 30 days

HEALTHY GROUP:

Inclusion Criteria:

* Absence of Parkinson's disease
* Mentally and physically capable to give informed consent

ALL SUBJECTS:

Exclusion Criteria:

* Atypical parkinsonian syndrome
* Cognitive impairment (MMSE ≥ 26)
* History of cerebro-vascular disease, epilepsy, or other disabling neurological diseases
* Psychiatric disorders, excepting mild depression (BDI score <14)
* Alcohol abuse
* Other clinically significant severe concomitant disease states
* Inability to follow the procedures of the study (e.g. due to language problems, psychological disorders, etc.)
* Participation in another study with investigational drug within the 60 days preceding and during the present project.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients with mild to moderate idiopathic Parkinson's Disease
  Control group (n=30): age-and sex-matched healthy volunteers, matched with the first 30 subjects with Parkinson's Disease enrolled in the study and with a complete dataset available.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Objective prospective and repeated assessment of motor function | from day 0 to day 15
  Finger tapping test

SECONDARY OUTCOMES:
Objective prospective and repeated assessment of motor function | from day 0 to day 15
  Tri-axial accelerometry (from wrist actigraphy)
Subjective prospective and repeated assessment of motor function | from day 0 to day 15
  Visual analogue scale (VAS)
Objective prospective assessment of sleep and wakefulness | from day 0 to day 15
  Wrist actigraphy
Subjective prospective assessment of sleep and wakefulness | from day 0 to day 15
  Electronic sleep diary
Subjective prospective assessment of sleepiness | from day 0 to day 15
  Stanford Sleepiness Scale (SSS)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Luca Ratti, MD, PhD, Principal Investigator — Neurocenter of Southern Switzerland
Locations (1):
- Sleep and Epilepsy center Department of Neurology, Neurocenter of Southern Switzerland, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Cock VC, Vidailhet M, Leu S, Texeira A, Apartis E, Elbaz A, Roze E, Willer JC, Derenne JP, Agid Y, Arnulf I. Restoration of normal motor control in Parkinson's disease during REM sleep. Brain. 2007 Feb;130(Pt 2):450-6. doi: 10.1093/brain/awl363. PMID 17235126
- [Background] Stefani A, Galati S, Peppe A, Bassi A, Pierantozzi M, Hainsworth AH, Bernardi G, Orlacchio A, Stanzione P, Mazzone P. Spontaneous sleep modulates the firing pattern of parkinsonian subthalamic nucleus. Exp Brain Res. 2006 Jan;168(1-2):277-80. doi: 10.1007/s00221-005-0175-y. Epub 2005 Nov 18. PMID 16328297
- [Background] Urrestarazu E, Iriarte J, Alegre M, Clavero P, Rodriguez-Oroz MC, Guridi J, Obeso JA, Artieda J. Beta activity in the subthalamic nucleus during sleep in patients with Parkinson's disease. Mov Disord. 2009 Jan 30;24(2):254-60. doi: 10.1002/mds.22351. PMID 18951542
- [Background] van Gilst MM, Bloem BR, Overeem S. "Sleep benefit" in Parkinson's disease: a systematic review. Parkinsonism Relat Disord. 2013 Jul;19(7):654-9. doi: 10.1016/j.parkreldis.2013.03.014. Epub 2013 Apr 21. PMID 23615667
- [Background] Merello M, Hughes A, Colosimo C, Hoffman M, Starkstein S, Leiguarda R. Sleep benefit in Parkinson's disease. Mov Disord. 1997 Jul;12(4):506-8. doi: 10.1002/mds.870120405. PMID 9251067
- [Background] Currie LJ, Bennett JP Jr, Harrison MB, Trugman JM, Wooten GF. Clinical correlates of sleep benefit in Parkinson's disease. Neurology. 1997 Apr;48(4):1115-7. doi: 10.1212/wnl.48.4.1115. PMID 9109914
- [Background] Tandberg E, Larsen JP, Karlsen K. Excessive daytime sleepiness and sleep benefit in Parkinson's disease: a community-based study. Mov Disord. 1999 Nov;14(6):922-7. doi: 10.1002/1531-8257(199911)14:63.0.co;2-7. PMID 10584665
- [Background] Bateman DE, Levett K, Marsden CD. Sleep benefit in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1999 Sep;67(3):384-5. doi: 10.1136/jnnp.67.3.384. No abstract available. PMID 10449564
- [Background] Sherif E, Valko PO, Overeem S, Baumann CR. Sleep benefit in Parkinson's disease is associated with short sleep times. Parkinsonism Relat Disord. 2014 Jan;20(1):116-8. doi: 10.1016/j.parkreldis.2013.09.005. Epub 2013 Sep 12. PMID 24084381
- [Background] Hogl BE, Gomez-Arevalo G, Garcia S, Scipioni O, Rubio M, Blanco M, Gershanik OS. A clinical, pharmacologic, and polysomnographic study of sleep benefit in Parkinson's disease. Neurology. 1998 May;50(5):1332-9. doi: 10.1212/wnl.50.5.1332. PMID 9595983
- [Background] Hogl B, Peralta C, Wetter TC, Gershanik O, Trenkwalder C. Effect of sleep deprivation on motor performance in patients with Parkinson's disease. Mov Disord. 2001 Jul;16(4):616-21. doi: 10.1002/mds.1138. PMID 11481684
- [Background] Hogl B, Gershanik O. Sleep benefit in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jun;68(6):798-9. doi: 10.1136/jnnp.68.6.798a. No abstract available. PMID 10877630
- [Background] Factor SA, Weiner WJ. 'Sleep benefit' in Parkinson's disease. Neurology. 1998 May;50(5):1514-5. doi: 10.1212/wnl.50.5.1514-b. No abstract available. PMID 9596032
- [Background] Noyce AJ, Nagy A, Acharya S, Hadavi S, Bestwick JP, Fearnley J, Lees AJ, Giovannoni G. Bradykinesia-akinesia incoordination test: validating an online keyboard test of upper limb function. PLoS One. 2014 Apr 29;9(4):e96260. doi: 10.1371/journal.pone.0096260. eCollection 2014. PMID 24781810
- [Derived] Mascheroni A, Choe EK, Luo Y, Marazza M, Ferlito C, Caverzasio S, Mezzanotte F, Kaelin-Lang A, Faraci F, Puiatti A, Ratti PL. The SleepFit Tablet Application for Home-Based Clinical Data Collection in Parkinson Disease: User-Centric Development and Usability Study. JMIR Mhealth Uhealth. 2021 Jun 8;9(6):e16304. doi: 10.2196/16304. PMID 34100767